CLINICAL TRIAL: NCT02943512
Title: Same Day Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alexandru Costea, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-3696
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Discharge day of Procedure (Experimental): Subjects in this arm will be discharged the same day of their cardiac device implant if deemed safe by treating physician.
  Interventions: Other: Discharge day of procedure
- Control (No Intervention): Subjects in this arm will remain in the hospital overnight per standard of care and will be discharged the next day if deemed safe by treating physician.

INTERVENTIONS:
Other: Discharge day of procedure — Subjects will be discharged the day of the procedure if safe
  Arms: Discharge day of Procedure

SUMMARY:
This study is to assess if subjects receiving a clinically indicated implanted cardiac pacemaker or defibrillator can be safely discharge home the same day of the procedure.

DETAILED DESCRIPTION:
Subjects who are implanted with a clinically indicated implanted cardiac pacemaker or defibrillator will be randomized to standard of care (next day discharge) versus same day discharge post implant. Both groups will under go standard of care assessments prior to discharge. The same day discharge group will receive a phone call the next day to assess for events and will transmit device data electronically. Both groups will be seen 10 - 14 days after implant for further evaluation.

The subjects will also complete questionnaires regarding their knowledge of self care and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for clinically indicated implant of cardiac pacemaker or defibrillator
2. Willing and able to provide informed consent
3. Appropriate clinical indication for the purpose of this study

   1. Primary prevention implantable cardioverter-defibrillator implant indicated for sudden cardiac death with ejection fraction more than 20%
   2. Sick sinus syndrome, non-high degree heart block as indication for pacemaker implant.
   3. No history of syncope
   4. No documented sudden cardiac death or ventricular arrhythmias requiring shock
4. Adequate social support to be able to comply with protocol.
5. Ability to complete remote monitor transmission

Exclusion Criteria:

1. Determined to be at risk for bleeding or on oral anticoagulation 2. Planned to be implanted with non-Biotronik device 3. Complete heart block as indication for permanent pacemaker 4. Secondary ICD indication 5. Immediate procedural complication requiring prolonged admission such as: pneumothorax, large hematoma, tamponade) determined during the procedure or immediately before discharge.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Average number of late complications between the 2 arms | up to 2 weeks after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Costea, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided